CLINICAL TRIAL: NCT02045303
Title: Healing Rate of Chronic and Sub-Acute Lower Extremity Ulcers Treated With Contact Ultrasound Followed by MIST Therapy: The VIP Ultrasound Protocol
Brief Title: Healing Rate of Leg Wounds Treated With Contact and Noncontact Ultrasound: The VIP Ultrasound Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Health Resources (Other)
Collaborators: Celleration, Inc. (Industry)
Responsible Party: Principal Investigator, Lisley Viana, Physical Therapist, Texas Health Resources
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004597
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Chronic Ulcer of Lower Extremity
Keywords: Sub-acute wound; Chronic wound; Wound; MIST; Soring; Contact Ultrasound; Noncontact ultrasound; Wound Care; VIP Ultrasound Protocol; Ultrasound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ambulatory Wound Clinic (Experimental): Intervention with contact ultrasound therapy and noncontact ultrasound therapy following the study protocol on subjects receiving care at the wound clinic.
  Interventions: Device: Contact Ultrasound Therapy; Device: Noncontact Ultrasound Therapy

INTERVENTIONS:
Device: Contact Ultrasound Therapy — Following our protocol, the ultrasound wound therapy will start with contact ultrasound until it meets criteria to switch to noncontact ultrasound therapy.
  Other Names: Soring, Sonoca-180
Device: Noncontact Ultrasound Therapy — Transition from contact to noncontact ultrasound when criteria for transition is met per our protocol.
  Other Names: Celleration Inc, MIST Therapy

SUMMARY:
Wound healing rate is higher when contact ultrasound therapy is followed by noncontact ultrasound therapy on sub-acute and chronic lower extremity ulcers of various etiologies requiring selective debridement, as compared to either Sonoca-180 or MIST Therapy alone.

DETAILED DESCRIPTION:
This prospective pilot study is designed to evaluate the clinical effectiveness of a wound care ultrasound treatment protocol for sub-acute or chronic wounds of the lower extremity and of any etiology. The Viana-Pompeo (VIP) ultrasound protocol consists of high intensity, low frequency, contact ultrasound therapy (with Sonoca-180) followed by low intensity, low-frequency, noncontact ultrasound therapy (with MIST Therapy). Previously published healing rates for each of the ultrasonic therapy modalities will be used as a comparison.

The Physical Therapist will perform the initial assessment and treatment, and devise an individualized plan of care that involves contact ultrasound followed by noncontact ultrasound. Subjects may remain in the study for up to 12 weeks, or up to when end of study criteria is met.

Transition from contact mode to noncontact mode will happen when:

- Wound is sufficiently clean with ≤ 20% of necrotic tissue or adherent slough.

OR

- >= 80% of soft slough is easily removed from the wound bed with mechanical or selective debridement before or after treatment

OR

- Wound bed quality has failed to progress after 3 consecutive contact ultrasound treatments

For the purposes of this study, treatments will be performed 3 times a week. Treatment time will be dependent on the wound area, at least 20 sec/cm2, per standard protocol.

Only the wounds present during Physical Therapy (PT) initial assessment will be included in the research. If the patient develops new wounds during the course of the research, the patient will receive appropriate treatment, but such wounds will not be part of the study.

Patients in the wound clinic setting are allowed to perform home dressing changes as ordered by the physician in addition to the dressing changes performed by the therapist or wound clinic nurse on clinic visit days. Patients and/or caregivers will be trained in dressing changes techniques and must understand the procedure prior to performing dressing changes on their own.

In addition to ultrasonic treatment and dressing changes, wound debridement may be performed each visit as needed. Digital photography and wound measurements will also be performed weekly and as needed.

End of PT wound therapy may be before, at, or after the end of the study period. The beginning of the MIST therapy will depend on the individual characteristics and wound needs.

A minimum of 4 MIST treatments must be completed for a patient's data to be included the data analysis in the acute care setting.

A minimum of 2 treatments per week (goal of 3 per week) must be reached for the 12 week period for a patient's data to be included in the data analysis.

Study Endpoints

Primary endpoint:

* Wound area reduction
* Percent granulation tissue
* Length of the study for ambulatory subjects: 12 weeks from Start of Contact Ultrasound therapy

Secondary endpoint:

* Wound closure at any point within the length of study
* Failure to note improvement in wound area, and/or wound volume, and/or wound bed quality after 4 consecutive weeks of treatment.
* 3 consecutive missed visits, or a total of 7 missed visits

ELIGIBILITY:
Inclusion Criteria:

* Patient is referred to Physical Therapy for contact ultrasound (which is included in the VIP protocol);
* Lower extremity (including foot) wound(s) of any etiology;
* Wound(s) presenting with slough, necrotic tissue, and/or non-viable tissue requiring debridement;
* Wound is present for 4 weeks or longer at the start of ultrasonic therapy;
* Insurance approval is obtained for Contact and Noncontact ultrasound treatments, in the ambulatory setting;
* Patient is 18 years of age or older;
* Female patient attesting not to be pregnant;
* Not undergoing Vacuum Assisted Closure (VAC) therapy.

Exclusion Criteria:

* Patient is referred to Physical Therapy for noncontact ultrasound only;
* Wound(s) not on lower extremity;
* Clean wound(s) that do not require debridement;
* Wound onset less than 4 weeks prior to the start of ultrasonic therapy;
* Malignancies on the treatment area;
* Patients in the ambulatory setting whose insurance did not approve them for both contact and noncontact ultrasound therapy;
* Patient is under 18 years of age;
* Female patient attesting to be pregnant;
* VAC Therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisley Viana, PTMS, Principal Investigator — Texas Health Resources - Presbyterian Hospital of Dallas
Locations (1):
- Texas Health Resources - Presbyterian Hospital of Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled subjects who had sub-acute or chronic lower leg wound requiring debridement, who were coming to the outpatient wound care clinic for follow up with wound care doctor.
Pre-assignment Details: The wound care doctor wrote orders for ultrasound therapy performed by Physical Therapist (PT). Throughout the open enrollment phase, the PT screened referred patients to check if they met study criteria.
Units Other Than Participants: Wounds
Groups:
- Ambulatory Wound Clinic - Wound Age Between 4 and 21 Weeks: Intervention with contact ultrasound therapy and noncontact ultrasound therapy following the study protocol on subjects receiving care at the wound clinic.
  Contact Ultrasound Therapy: Following our protocol, the ultrasound wound therapy will start with contact ultrasound until it meets criteria to switch to noncontact ultrasound therapy.
  Noncontact Ultrasound Therapy: Transition from contact to noncontact ultrasound when criteria for transition is met per our protocol.
  Wound age between 4 and 21 weeks
- Ambulatory Wound Clinic - Wound Age Between 22 and 46 Weeks: Intervention with contact ultrasound therapy and noncontact ultrasound therapy following the study protocol on subjects receiving care at the wound clinic.
  Contact Ultrasound Therapy: Following our protocol, the ultrasound wound therapy will start with contact ultrasound until it meets criteria to switch to noncontact ultrasound therapy.
  Noncontact Ultrasound Therapy: Transition from contact to noncontact ultrasound when criteria for transition is met per our protocol.
  Wound age between 22 and 46 weeks
- Ambulatory Wound Clinic - Wound Age >= 47 Weeks: Intervention with contact ultrasound therapy and noncontact ultrasound therapy following the study protocol on subjects receiving care at the wound clinic.
  Contact Ultrasound Therapy: Following our protocol, the ultrasound wound therapy will start with contact ultrasound until it meets criteria to switch to noncontact ultrasound therapy.
  Noncontact Ultrasound Therapy: Transition from contact to noncontact ultrasound when criteria for transition is met per our protocol.
  Wound age >= 47 weeks
Period: Overall Study
Arm/Group | Ambulatory Wound Clinic - Wound Age Between 4 and 21 Weeks | Ambulatory Wound Clinic - Wound Age Between 22 and 46 Weeks | Ambulatory Wound Clinic - Wound Age >= 47 Weeks
Started | 6; 6 Wounds | 3; 10 Wounds | 2; 8 Wounds
Completed | 4; 4 Wounds | 0; 0 Wounds | 2; 8 Wounds
Not Completed | 2; 2 Wounds | 3; 10 Wounds | 0; 0 Wounds
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Wounds
Groups:
- Wound Age Between 4 and 21 Weeks: Both groups underwent the same protocol of contact ultrasound followed by non-contact ultrasound therapy, with the goal of 3x/week treatment frequency. Study data for this group was collected over a period of 12 weeks or up to the time of wound closure.
- Wound Age >=47 Weeks: Both groups underwent the same protocol of contact ultrasound followed by non-contact ultrasound therapy, with the goal of 3x/week treatment frequency. Study data for this group was collected over a period of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Wound Age Between 4 and 21 Weeks | Wound Age >=47 Weeks | Total
Number analyzed (Participants) | 4 | 2 | 6
Number analyzed (Wounds) | 4 | 8 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0
  Black | 1 | 1 | 2
  Hispanic or Latino | 0 | 0 | 0
  White | 3 | 1 | 4
Wound Location [Count of Units; unit: Wounds]
  Ankle | 0 | 1 | 1
  Foot/Heel/Toes | 3 | 2 | 5
  Knee | 0 | 1 | 1
  Lower Leg | 1 | 4 | 5
Initial Wound Area [Mean (Full Range); unit: cm^2] | 10.12 [1.92 to 15.36] | 7.93125 [1.02 to 18.6] | 8.66083 [1.02 to 18.6]
Associated Diagnosis [Count of Units; unit: Wounds]
  S/p Ganglion Cyst Removal | 1 | 0 | 1
  Stage IV Pressure Ulcer | 1 | 0 | 1
  Diabetes | 2 | 3 | 5
  Peripheral Artery Disease | 2 | 0 | 2
  Above Knee Amputation (opposite limb) | 1 | 0 | 1
  Post-Surgical Debridement | 1 | 0 | 1
  Vasculitis | 0 | 3 | 3
  Cat Bite | 1 | 0 | 1
  3rd Degree Burn | 0 | 5 | 5
  Venous Insufficiency | 0 | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Total Wound Area
Description: Mean and Standard Deviation of the group's total wound area at day one and last treatment day. Wound area was measured as Length x Width. This is to assess the change in area, in order to assess wound progress towards closure.
Time Frame: Initial measurement at day 1 and measurement at the subject's last visit at 12 weeks or sooner if the wound closed before then.
Measure: Mean (Standard Deviation); unit: Squared centimiters
Units Other Than Participants: Wounds
Groups:
- Wound Age Between 4 and 21 Weeks: Wounds age between 4 and 21 weeks at the day of initial visit.
- Wound Age >=47 Weeks: Wounds age >=47 weeks at the day of initial visit.
Arm/Group | Wound Age Between 4 and 21 Weeks | Wound Age >=47 Weeks
Number analyzed (Participants) | 4 | 2
Number analyzed (Wounds) | 4 | 8
Squared centimiters
  Initial Wound Area | 7.93125 (5.96128) | 7.93125 (5.96128)
  Wound Area on Last Study Visit | 1.3275 (2.61515) | 8.80875 (7.73304)

2. Secondary Outcome: Total Wound Volume
Description: Mean and Standard Deviation of the group's total wound volume at day one and last treatment day. Wound volume was measured as Length x Width X Depth (when able to determine depth). This is to assess the change in volume, in order to assess wound progress towards closure.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: cubic centimeter
Units Other Than Participants: Wounds
Groups:
- Wound Age Between 4 and 21 Weeks: Wounds with age between 4 and 21 weeks at the day of initial visit.
- Wound Age >=47 Weeks: Wounds with age >= 47 weeks at the day of initial visit.
Arm/Group | Wound Age Between 4 and 21 Weeks | Wound Age >=47 Weeks
Number analyzed (Participants) | 4 | 2
Number analyzed (Wounds) | 4 | 8
cubic centimeter
  Initial Wound Volume | 9.561 (9.94704) | 2.67475 (2.73782)
  Wound Volume on Last Study Visit | 0.394 (0.78401) | 2.086 (1.9324)

3. Secondary Outcome: Wounds With Slough/Eschar Reduction on Visit 2 and Wounds With Slough/Eschar Reduction at Last Visit
Description: Mean and Standard Deviation of the group's percent adherent and/or non-adherent slough present in the wound bed at day one and last treatment day. This is to assess the change in slough/eschar. This is to determine progression from contact to noncontact ultrasound therapy, as well as to determine progress of wound bed quality.
Time Frame: Day 2 and measurement at the subject's last visit at 12 weeks or sooner if the wound closed before then.
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Groups:
- Wound Age >=47 Weeks: Wounds age between >=47 weeks at the day of initial visit.
Arm/Group | Wound Age Between 4 and 21 Weeks | Wound Age >=47 Weeks
Number analyzed (Participants) | 4 | 2
Number analyzed (Wounds) | 4 | 8
Wounds
  Wounds w/ slough/eschar Reduction on visit 2 | 4 | 8
  Wounds w/ slough/eschar Reduction on last visit | 4 | 7

4. Other Pre Specified Outcome: Wounds With Granulation Present on Visit 1 and Wounds With Granulation Present at Last Visit
Description: Mean and Standard Deviation of the group's total percent of granulation tissue present in the wound bed at day one and last treatment day. This is to assess the change in granulation, in order to assess progress of wound bed quality.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: % Granulation
Units Other Than Participants: Wounds
Arm/Group | Wound Age Between 4 and 21 Weeks | Wound Age >=47 Weeks
Number analyzed (Participants) | 4 | 2
Number analyzed (Wounds) | 4 | 8
% Granulation
  Initial Granulation | 22.5 (17.07825) | 21.75 (24.97284)
  Granulation on last visit | 100 (0) | 55.125 (38.93745)

ADVERSE EVENTS:
Time Frame: Therapist was monitoring for adverse effects on subjects on both study arms throughout the study duration (12 weeks) and for the duration of the therapy (if the subject continued therapy passed the 12 weeks), but no adverse events were observed, therefore no data was collected.
Groups:
- Wound Age Between 4 and 21 Weeks: Wounds age between 4 and 21 weeks
- Wound Age >=47 Weeks: Wounds age equal to or greater than 47 weeks
Arm/Group | Wound Age Between 4 and 21 Weeks | Wound Age >=47 Weeks
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes